CLINICAL TRIAL: NCT06196099
Title: Combining Resting Blood Flow Restriction with Neuromuscular Electrical Stimulation: Effects on Blood Lactate Levels and Lower Limb Muscle Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hyunjoong Kim (Other)
Responsible Party: Sponsor-Investigator, Hyunjoong Kim, Investigator, Sahmyook University
Organization: Sahmyook University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1041223-202309-HR-30
Record Dates: First submitted 2023-12-23; First posted 2024-01-09 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- rest-Blood Flow Restriction plus Neuromuscular Electrical Stimulation (Active Comparator)
  Interventions: Device: Blood Flow Restriction; Device: Neuromuscular Electrical Stimulation
- rest-Blood Flow Restriction (Active Comparator)
  Interventions: Device: Blood Flow Restriction
- Squat Exercise (Active Comparator)
  Interventions: Behavioral: Squat exercise

INTERVENTIONS:
Device: Blood Flow Restriction — The study participants were instructed to rest quietly in a seated position for 10 minutes. During the last 3 minutes of the resting period, upper arm blood pressure was measured twice using an automatic blood pressure monitor (BP170, InBody, Korea). The blood flow restriction cuffs (BFR Therapy Cuff, BFR Therapy Co., USA) - measuring 5cm in width and 60cm in length - were applied to the upper third of the thigh on both legs. To maintain consistency in measurements, the distance from the proximal part of the kneecap to the distal edge of the cuff was measured. A Capillary Reaction Time (CRT) test was used to assess the appropriateness of the cuff pressure; this involved applying thumb pressure to the quadriceps muscle after cuff application and timing how long it took for the skin color to return to normal.
  Arms: rest-Blood Flow Restriction; rest-Blood Flow Restriction plus Neuromuscular Electrical Stimulation
Device: Neuromuscular Electrical Stimulation — Neuromuscular Electrical Stimulation (NMES) was applied five times a week for one week using a four-channel stimulator (Compex Physio, Chattanooga, Switzerland). The stimulation protocol was set to a frequency of 35Hz, with electrodes attached to the vastus lateralis and vastus medialis muscles. The therapist adjusted the intensity and alternating output of the electrodes selectively to facilitate the squat exercises required during the intervention. During the stimulation period, participants were engaged in a squat exercise program, with the total duration of stimulation being 10 minutes.
  Arms: rest-Blood Flow Restriction plus Neuromuscular Electrical Stimulation
Behavioral: Squat exercise — In this study, the squat exercise was performed in four sets. Participants were instructed to position their feet shoulder-width apart and educated to squat in such a way that their knees did not extend beyond their toes. To ensure consistency in performing the squat at the same angle, a mark was made on the wall at the pelvic height during a 90° squat. This allowed participants to perform squats at the same height. The exercise was conducted under the guidance of a physical therapist with five years of clinical experience.
  Arms: Squat Exercise

SUMMARY:
The current research landscape shows studies indicating increased muscle strength and hypertrophy through neuromuscular electrical stimulation combined with blood flow restriction. However, there is a lack of research specifically on the effects of this combination during rest periods. Therefore, the primary objective of this study is to investigate the impact of resting blood flow restriction training combined with neuromuscular electrical stimulation on blood lactate levels and changes in lower limb muscle function in healthy male adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males in their 20s,
* Individuals who answered less than one item on the PAR-Q (Physical Activity Readiness Questionnaire),
* Participants who consented to the use and publication of their physical function evaluation data and expressed a desire to participate in the exercise experiment.

Exclusion Criteria:

* Individuals with severe hypertension (blood pressure above 170/110 mmHg),
* Individuals with a history of deep venous thrombosis,
* Individuals with endothelial dysfunction,
* Individuals with peripheral vascular disease,
* Individuals with one or more of the following conditions: diabetes, infection, cancer,
* Participants who expressed a desire to withdraw during the study period or whose participation rate was below 80% were excluded from the study.

Ages: 20 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Blood lactate | Immediate change from baseline after intervention
  Lactate levels were measured using the Accutrend Plus (Roche, Germany). A small amount of whole blood was collected from the participants for blood lactate concentration analysis. The procedure involved the finger-prick method, where the tip of the right index finger was disinfected with an alcohol swab. Then, a lancet prepared for this purpose was used to obtain a small sample of capillary blood from the disinfected area. The collected blood was then applied to lactate strips, and the blood lactate analyzer (Accutrend Plus, Roche, Germany) provided the lactate level readings within 60 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Honam University, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: Yes